CLINICAL TRIAL: NCT04602091
Title: JAKINIB Study: " 'Observational', Multicentre Trial Collecting Prospective and On-going Clinical and Laboratory Data for Patients Treated With JAK Inhibitors for Inflammatory Rheumatism According to EMA."
Brief Title: Observational Study in Patients Treated With JAK Inhibitors for Inflammatory Rheumatism (MAJIK)
Acronym: MAJIK
Status: Active, not recruiting | Type: Observational
Sponsor: Societe Francaise de Rhumatologie (Other)
Collaborators: Bordeaux PharmacoEpi (Other)
Responsible Party: Sponsor
Other Study IDs: MAJIK Registry
Record Dates: First submitted 2020-10-14; First posted 2020-10-26 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Rheumatoid Arthritis; Inflammatory Rheumatism; Psoriatic Arthritis; Spondyloarthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Rheumatic Fever; Arthritis, Psoriatic; Spondylarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | US Export: No

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Janus kinase (JAK) inhibitors are a new class of molecules available to the therapeutic arsenal for chronic inflammatory rheumatic diseases.The tolerance profile of this new class needs to be better defined and its use in real life further established.

The French Society of Rheumatologists intends to coordinate a prospective national registry study for this follow-up.

This registry will include at least 1500 Rheumatoid Arthritis (RA) and 150 patients with psoriatic arthritis from the start of treatment with JAK inhibitor and then followed for 5 years.

This registry is a longitudinal, multicentre, observational registry study. The objective of this national registry is to get a better understanding of the safety profiles of JAK inhibitors and get knowledge of their use in daily practice in order to optimize this use and potentially integrate JAK inhibitors into personalised medicine strategies.

This registry will generate efficacy data, especially therapeutic maintenance, observation, allowing inter-registry comparisons with other biologic compounds in the French population, and can be aggregated with other similar registries in other countries.

DETAILED DESCRIPTION:
Design:

This registry is a longitudinal, multicentre, observational registry study, with continuous and ambispective collection of clinical and laboratory data. The patients will be followed for 5 years, regardless of the therapeutic modifications occurring thereafter.

Target population:

Patients initiating JAK inhibitor therapy for inflammatory rheumatic disorder.

Number of patients and centres :

* The objective is to include, per drug available on the market, at least 300 to 500 patients with RA and at least 100 to 150 patients with psoriatic arthritis. If a JAK inhibitor is approved in a new indication of chronic rheumatic disease by European Medicines Agency (EMA), the number of patients to include for each molecule in this indication will be adjusted as a function of the prevalence/epidemiology of each disease. Products currently available (baricitinib and tofacitinib) will be considered at the start of this registry; then every new indication for an already approved drug or every new drug in the same therapeutic class starting from the date they are placed on the market will be considered.
* More than 80 centers in France (hospital-based, public and private practice) will participate.

ELIGIBILITY:
Inclusion criteria

* Patients older than 18
* Patient treated with a JAK inhibitor in accordance with EMA, for chronic inflammatory rheumatisms, independent of the therapeutic line
* Subject who is a member of a social security regime
* Free, declared, written consent signed by the subject and the investigator on the day of inclusion Exclusion criteria
* Patient who cannot understand the implications and rules of the study
* Patient opposition to participating in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: French patients treated for chronic inflammatory rheumatic disorders according to EMA.
Sampling Method: Non-Probability Sample
Enrollment: 2300 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Therapeutic maintenance of JAK inhibitors | From the beginning of the study up to Year 1
  The therapeutic maintenance will be measured by the retention rate ie the percentage of patients remaining treated by JAK inhibitors.

SECONDARY OUTCOMES:
Real-life tolerance of JAK inhibitors | From the beginning of the study until the end of the 5 years follow-up
  Occurence of adverse events and action taken (temporary or final stop to JAK inhibitor treatment upon the occurrence of adverse event).
Real-life tolerance of JAK inhibitors in sub-groups | From the beginning of the study until the end of the 5 years follow-up
  Occurence of adverse events and action taken (temporary or final stop to JAK inhibitor treatment upon the occurrence of adverse event), in an older population or presenting with comorbidities
Efficacy of JAK inhibitors | From the beginning of the study until the end of the 5 years follow-up
  Evaluated using clinical data (list is not exhaustive): number of swelling joints (NAG), number of tender joints (NAD), erythrocyte sedimentation rate (ESR), levels of C-reactive protein (CRP), the visual analogic scale (VAS) for disease activity evaluated by the patient and by the physician.
Comparison of JAK inhibitors efficacy (monotherapy versus combination with DMARDS) | From the beginning of the study until the end of the 5 years follow-up
  Evaluate the efficacy of JAK inhibitors administered as monotherapy versus combination with a conventional synthetic DMARDs
Efficacy of JAK inhibitors dose (full doses versus half doses) | From the beginning of the study until the end of the 5 years follow-up
Use of JAK inhibitors in current practice | From the beginning of the study until the end of the 5 years follow-up
  Starting dosage, therapeutic adjustments, etc.
Place of JAK inhibitors in real-life practice in the treatment arsenal for patients with chronic inflammatory rheumatic disorders | From the beginning of the study until the end of the 5 years follow-up
  Therapeutic history of the patient regarding DMARDs before starting treatment with a JAK inhibitor
Patient reported outcomes: Quality of life | From the beginning of the study until the end of the 5 years follow-up
  Analyse the effect of JAK inhibitors on patient reported outcomes in regard to quality of life and functional impact : Health Assessment Questionnaire (HAQ) questionnaire
Patient reported outcomes: Acceptance | From the beginning of the study until the end of the 5 years follow-up
  Analyse the effect of JAK inhibitors on patient reported outcomes in regard to acceptance : treatment acceptance questionnaire
Patient reported outcomes: Compliance | From the beginning of the study until the end of the 5 years follow-up
  Analyse the effect of JAK inhibitors on patient reported outcomes in regard to Compliance : compliance questionnaire (Morisky-Green self-questionnaire)
Drug interactions | From the beginning of the study until the end of the 5 years follow-up
  Identify new drug interactions
Analysis if data from a National Health Database (SNIIRAM): demographics | From the beginning of the study until the end of the 5 years follow-up
  With and without chaining to the patients included in this cohort with the possibility of evaluating demographics
Analysis if data from a National Health Database (SNIIRAM): medical economics | From the beginning of the study until the end of the 5 years follow-up
  With and without chaining to the patients included in this cohort with the possibility of evaluating medical economics
Analysis if data from a National Health Database (SNIIRAM): compliance | From the beginning of the study until the end of the 5 years follow-up
  With and without chaining to the patients included in this cohort with the possibility of evaluating compliance
Establishment of an open database | From the beginning of the study until the end of the 5 years follow-up
  Establish an open database which can be integrated with other national registries with a view toward future international analyses

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Elise TRUCHETET, Principal Investigator — CHU de Bordeaux - Pellegrin; Jerôme AVOUAC, Principal Investigator — AP-HP Hôpital Cochin; Clément PRATI, Principal Investigator — CHRU de Besançon
Locations (60):
- France (60):
  - CH Antibes, Antibes
  - Private office, Bayonne
  - CH Franche Comte, Belfort
  - CHU de Besançon, Besançon
  - AP-HP Avicenne, Bobigny
  - CHU de Bordeaux, Bordeaux
  - CH Bourg-en-Bresse, Bourg-en-Bresse
  - CHRU Brest, Brest
  - CHU Caen, Caen
  - CH Cannes, Cannes
  - CH Chartres, Chartres
  - CH Cholet, Cholet
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CH Colombes, Colombes
  - AP-HP Henri Mondor, Créteil
  - CH Dax, Dax
  - CH de Dijon, Dijon
  - CH de Douai, Douai
  - CHD de Vendee, La Roche-sur-Yon
  - CH La Rochelle, La Rochelle
  - CHG Jacques Monod, Le Havre
  - AP-HP Bicetre, Le Kremlin-Bicêtre
  - CH Le Mans, Le Mans
  - CHU Lille, Lille
  - Private office, Limoges
  - CH Saint Philibert, Lomme
  - CHU Lyon, Lyon
  - Infirmerie protestante de Lyon, Lyon
  - CHU Marseille Sainte-Marguerite, Marseille
  - Hôpital Saint Joseph, Marseille
  - CH Mont de Marsan, Mont-de-Marsan
  - CHU de Montpellier, Montpellier
  - CH Morlaix, Morlaix
  - GH de Mulhouse, Mulhouse
  - CHU Nantes, Nantes
  - CH Nevers, Nevers
  - CHU Nice, Nice
  - CH Niort, Niort
  - CH Orleans, Orléans
  - AP-HP Ambroise Pare, Paris
  - AP-HP Bichat, Paris
  - AP-HP Lariboisiere, Paris
  - AP-HP Pitie-Salpetriere, Paris
  - AP-HP Saint Antoine, Paris
  - Hopital La Croix Saint Simon, Paris
  - Hôpital Cochin, Paris
  - CH Pau, Pau
  - CHU Reims, Reims
  - CHU Rouen, Rouen
  - CHU de la Reunion, Saint-Denis
  - CHU Saint Etienne, Saint-Etienne
  - CH Bégin, Saint-Mandé
  - CH Saint Nazaire, Saint-Nazaire
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU Tours, Tours
  - CH Troyes, Troyes
  - CH Valence, Valence
  - CH Valenciennes, Valenciennes
  - Polyclinique Vauban, Valenciennes